CLINICAL TRIAL: NCT06286657
Title: Xanthohumol in the Prevention of Virus-mediated Upper Respiratory Tract Infections in Humans
Brief Title: Xanthohumol and Viral Infections (XL)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Vienna (Other)
Responsible Party: Principal Investigator, Prof. Dr. Ina Bergheim, Prof. Dr. Ina Bergheim, University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: UVienna23a
Record Dates: First submitted 2024-01-17; First posted 2024-02-29 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Infection Viral
MeSH Terms: conditions — Virus Diseases | interventions — xanthohumol

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): Participants consume twice per day a study drink which contains 0,75 mg soluble Xanthohumol for 90 days
  Interventions: Dietary Supplement: Xanthohumol
- Placebo (Experimental): Participants consume twice per day a study drink which contains 0 mg soluble Xanthohumol for 90 days
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Xanthohumol — Participants consume twice per day a study drink which contains 0,75 mg soluble Xanthohumol for 90 days
  Arms: Intervention
Dietary Supplement: Placebo — Participants consume twice per day a study drink which contains 0 mg soluble Xanthohumol for 90 days
  Arms: Placebo

SUMMARY:
The aim of the present study is to determine if a regular oral supplementation of xanthohumol attenuate the severity of symptoms and duration of´viral infections.

DETAILED DESCRIPTION:
In this placebo-controlled study, blood is taken on the first day of the study, followed by a 90-day intervention with xanthohumol or a placebo, which is taken twice daily. Blood samples will be taken on day 0, day 45 and day 90. Should the study participants develop a respiratory infection during the study, they will be asked to perform a self-test.

ELIGIBILITY:
Inclusion Criteria:

* healthy
* BMI >18 kg/m² or < 28kg/m²

Exclusion Criteria:

* food intolerances
* food allergies
* chronic inflammatory diseases
* metabolic diseases
* viral or bacterial infections within the last 3 weeks of inclusion
* intake of immunosuppressive medication
* severe acute respiratory syndrome coronavirus type 2-infection in the last 4 months
* influenza infection in the "current" flu season

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Changes in severity and duration of viral infections | 90 days
  Changes in score of Wisconsin Upper Respiratory Symptom Survey

SECONDARY OUTCOMES:
Changes in blood lipid levels | 90 days
  Changes in triglyceride levels (mg/dl) and cholesterol levels (mg/dl)
Changes in cognitive skills | 90 days
  Assessment of cognitive processes using stroop test

CONTACTS AND LOCATIONS:
Locations (1):
- University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No